CLINICAL TRIAL: NCT06566573
Title: Does the Degree of Stenosis Affect Cervical Proprioception in Patients With Cervical Problems?
Brief Title: Does the Degree of Cervical Stenosis Affect Proprioception?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Onur Engin, Assist.Prof., Izmir Democracy University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: cervicalproprioception35
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Proprioceptive Disorders; Stenosis
MeSH Terms: conditions — Somatosensory Disorders; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Prospective cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cervical stenosis degree 0 (Other): Pain, range of motion and proprioceptive sensations of patients with spinal stenosis grade 0 according to the Kang grading system will be evaluated on MRI.
  Interventions: Other: Pain; Other: Normal Range of Motion; Other: Proprioceptive Sense
- cervical stenosis degree 1 (Other): Pain, range of motion and proprioceptive sensations of patients with spinal stenosis grade 1 according to the Kang grading system will be evaluated on MRI.
  Interventions: Other: Pain; Other: Normal Range of Motion; Other: Proprioceptive Sense
- cervical stenosis degree 2 (Other): Pain, range of motion and proprioceptive sensations of patients with spinal stenosis grade 2 according to the Kang grading system will be evaluated on MRI.
  Interventions: Other: Pain; Other: Normal Range of Motion; Other: Proprioceptive Sense
- cervical stenosis degree 3 (Other): Pain, range of motion and proprioceptive sensations of patients with spinal stenosis grade 3 according to the Kang grading system will be evaluated on MRI.
  Interventions: Other: Pain; Other: Normal Range of Motion; Other: Proprioceptive Sense

INTERVENTIONS:
Other: Pain — The relationship between the degree of stenosis and pain in patients with lumbar spinal stenosis will be evaluated with a visual analogue scale.
Other: Normal Range of Motion — CROM will be used for normal range of motion (ROM) of the cervical region. Measurements will be made separately for flexion, extension, right rotation, left rotation, right and left lateral flexion.
Other: Proprioceptive Sense — CROM will be used for cervical proprioception. Measurements will be made separately for flexion, extension, right rotation, left rotation, right and left lateral flexion.

SUMMARY:
Neck pain is a common health problem that negatively affects the quality of life of individuals of different age groups and most people experience this problem at some point in their lives. With age, changes occur in the neuromuscular functions of the cervical region that are considered normal. These changes lead to many problems such as postural disorder, decreased stabilization, loss of normal joint motion, balance disorders and decreased cervical joint position sense. When the literature was examined, the situation was observed that cervical proprioception, which is defined as joint position sense, has not been sufficiently investigated. In particular, researchers have not found any literature on how proprioceptive sensation varies according to the degree of cervical stenosis. Therefore, this study will provide a direction for the treatment of cervical region problems. The data will be discussed with appropriate statistical methods and treatment recommendations will be presented according to the results obtained.

DETAILED DESCRIPTION:
With the increase in technology, the use of computers in the workplace is becoming widespread all over the world. With the use of computers in offices, long-term computer exposure of employees at the desk has emerged. In recent years, the use of computers is not only limited to offices, but the concept of working remotely from home is becoming increasingly widespread as a result of extraordinary conditions such as pandemics and earthquakes. Long-term work at the desk causes various musculoskeletal disorders. These musculoskeletal system disorders, which develop due to working life, were first mentioned by Bernardino Ramazini in the 17th century in his book "Occupational Diseases", including the pain in the hands of bakery workers and posture disorders of desk workers. Repetitive movements and static posture, use of wrong body mechanics and inadequate ergonomic conditions play a role in the development of musculoskeletal disorders in desk workers. In addition to these, stress experienced at work is also effective in musculoskeletal disorders. Neck pain is the most common complaint in desk workers. When neck musculoskeletal complaints are investigated, neck pain is seen in the first place with a high rate of 65.7%. In addition, it has been reported that 22% of the employees have head, neck and back pain in different parts of the individuals due to the high duration of time spent in sitting position.

Degenerative problems frequently occur in the cervical spine. Cervical spondylosis, cervical degenerative disc disease / disc herniation, cervical spondylotic myopathy conditions, which are frequently seen due to degeneration in the cervical spine, cause canal narrowing in the cervical region. Cervical spinal canal being narrower than normal is defined as cervical spinal stenosis. Cervical spinal stenosis causes a variety of symptoms depending on its severity. The most common symptom of cervical spinal stenosis is neck pain, which may be accompanied by stiffness and limited range of motion. Other symptoms may include abnormal reflexes in the upper limbs, cervical spine pain, nerve root compression in the cervical region, cervical cord compression, numbness or tingling in the arms, hands, legs or feet, weakness in the arms, hands, legs or feet, difficulty with coordination and balance, and in severe cases, loss of bladder or bowel control.

The diagnosis of cervical spinal stenosis is made by evaluating the patient's medical history, physical examination findings and imaging tests. Firstly, the patient's symptoms such as neck pain, numbness, weakness in arms and legs are questioned. Previous injuries and medical conditions that may cause symptoms are also questioned. In the physical examination, findings related to spinal cord compression such as abnormal reflexes or muscle weakness are evaluated. Other tests may also be performed to assess the patient's range of motion or the function of the spinal cord and nerve roots.

Imaging tests, such as magnetic resonance imaging (MRI) or computed tomography (CT) scans, can provide detailed images of the spine and help determine the location and severity of stenosis. In a study on the role of MRI in guiding the diagnosis and treatment of cervical spinal stenosis syndromes, it was found that there was an agreement between the clinical presentation of cervical canal stenosis and imaging findings.

Symptoms of cervical spinal stenosis are diverse and can include both sensory and motor impairments. A case study in the literature of a person with severe cervical spinal stenosis showed that the patient had difficulty walking, weakness in the right leg and unsteadiness in walking. Sensory examination revealed mild tactile pain and decreased proprioception. In addition, another study investigating the effectiveness of MRI in diagnosis and treatment showed that one of the most common symptoms in patients with cervical canal stenosis was the presence of abnormal reflexes in the tendons of the upper extremities. These studies show the potential effects of cervical spinal stenosis on proprioception.

Proprioception is used to describe the information amplified by afferent receptors towards the central nervous system (CNS) that contributes to the neuromuscular control of movement. This definition encompasses kinesthesia, the perception of joint movement, and joint position sense, the perception of joint position sensation. Spatial orientation is a key process required for many functions such as coordinating movement and maintaining posture. Sensorimotor control of head and eye movements in stable upright posture relies on afferent information from the vestibular, visual and proprioceptive systems that converge at various sites throughout the CNS. The cervical spine plays an important role in providing proprioceptive input and this is explained by the abundance of cervical mechanoreceptors and their central and reflex connections to the vestibular, visual and CNS.

Impaired proprioception has negative effects on motor control and muscle stiffness, which explains symptoms such as balance problems and clumsiness in musculoskeletal disorders. Decreased impulses to alpha motor neurons, impaired reflex joint stabilization, increased postural oscillation and increased errors in the visual component of movement are also associated with proprioception loss. In addition, dizziness, visual disturbances and changes in the control and coordination of head and eye movements are also observed in individuals with cervical proprioception loss. When loss of proprioception persists long-term, the pathophysiologic risk of injury increases due to impaired motor output from the CNS and inadequate muscular protection of joint tissue, leading to recurrence or persistence of pain disorders, including the onset and progression of secondary osteoarthrosis. Muscle performance is reduced due to impaired mechanoreceptor input to the CNS from injured tissues and this has been associated with the onset and progression of osteoarthrosis in peripheral joints. Cervical proprioception is impaired in relation to pain, effusion, trauma, fatigue and various musculoskeletal disorders.

Cervical proprioception impairment leading to cervical sensorimotor control disorders is one of the main problems in patients with neck pain. Cervical sensorimotor control involves central integration and processing of all afferent information including visual, vestibular and cervical proprioceptive inputs. In addition, the execution of the motor program through the cervical muscles contributes to maintaining head posture and balance, as well as the stability of the cervical joints. Although the importance of proprioception in other regional pains has been understood, there are not enough studies in the literature for the neck region. In their study, Reddy et al. found that proprioception sensation was impaired in patients with cervical pain and cervical spondylosis compared to the normal population.

In this study, CROM, which is a normal joint motion measurement device that will be used in this study, was used to evaluate cervical range of motion and proprioception.

Cervical disc disorders and cervical stenosis have an important place in the etiology of cervical pain. However, the relationship between the degree of cervical stenosis and the amount of impairment of proprioception sensation has not been examined in the literature. Therefore, this relationship will be examined in this study. It is thought that the data obtained in this study will be decisive in shaping the exercise program and directing the treatment in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Previously performed cervical MRI
* Cases whose stenosis classification can be clearly determined on MRI

Exclusion Criteria:

* Individuals who did not agree to participate in the study
* Individuals undergoing cervical surgery
* Those with pain that restricts cervical movement
* Those diagnosed with vertigo
* Those with sudden hearing loss
* Having additional neurological disorders
* Those with psychiatric and cognitive disorders that would prevent measurement in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | through study completion, an average of 1 year
  Visual analog scale (VAS) will be used for pain assessment. The VAS is a one-dimensional measure of pain intensity and is frequently used in adult populations. The pain definitions used for the two endpoints on a 10 cm line are 0 for 'no pain' and 10 for 'extreme pain. Pain will be evaluated in 3 different ways: pain at the time, pain at rest and pain during activity. While assessing pain, the type and location of pain will also be questioned verbally and noted.
Assessment of Normal Joint Motion | through study completion, an average of 1 year
  Normal range of motion (ROM) of the cervical region will be assessed with the Pa Crom Basic - Cervical Range Of Motion (CROM). CROM is an instrument that reliably measures cervical range of motion. The instrument is fixed to the patient's head with velcro. Patients sit in a chair and their feet are flat on the floor. The CROM dial is set to position 0 in the plane to be measured. Patients are shown how to perform the movement and are asked to actively perform this movement. Measurements are made separately for flexion, extension, right rotation, left rotation and right-left lateral flexion movements. Each movement is performed three times and passive range of motion is evaluated. The average of the test values is recorded.
Assessment of cervical proprioception | through study completion, an average of 1 year
  Cervical proprioception will be assessed with the CROM instrument. To test neck proprioception, the ability to reposition the head will be examined. It is assessed in two ways: 1. Repositioning to a neutral head position (Joint Position Error - EPH) 2. Repositioning the head to a predetermined reference point (Head Repositioning Accuracy - HRPA). For CBPD, the patient is asked to reposition the head to a predetermined target position; 2-2.5 degrees deviation is normal, 3-4 degrees deviation is impaired. The patient sits upright in a chair, the CROM device is fixed to the head with velcro. In EPH, the head is held in normal position with an eye patch and deviations in CROM are recorded. In BYPD, the head is positioned in the determined position with the eye patch closed and the amount of deviation is averaged. Measurements are made in flexion, extension, right and left rotation and lateral flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University; Ayşe Sezgi Kızılırmak Karataş, Msc. Pt., Principal Investigator — Izmir Democracy University